CLINICAL TRIAL: NCT04607018
Title: Effect of Panaceo Micro Activation (PMA)-Zeolite-Clinoptilolite on the Mineral Metabolism and Selected Blood Parameters (MMBP Study)
Brief Title: Effect PMA-Zeolite on the Mineral Metabolism and Blood Parameters (MMBP Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Pula (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMBP_study
Record Dates: First submitted 2020-05-18; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Effects of the Elements

STUDY DESIGN:
Intervention Model Description: The pilot-study evaluated the effect of the PMA-zeolite supplementation of 28 days (in accordance with the regulations of this medical device) on 2 groups of 15 subjects (males and females) all together. All subjects are healthy volunteers taking PMA-zeolite since years and the other one just started. No washout phase is planned, but if food-supplements are taken this will be protocolled. The diagnostics will be performed through the defined parameters at defined time-points.
Masking Description: no masking - all are taking the same products starting at different time points
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic intake group (Active Comparator): healthy subjects (control group) receive PMA-zeolite as powder. They take the product already before the study started (since 28 days before or even longer)
  Interventions: Device: PMA-zeolite
- Naive intake group (Active Comparator): healthy subjects (control group) receive PMA-zeolite as powder. They take the product only since the first day of the study
  Interventions: Device: PMA-zeolite

INTERVENTIONS:
Device: PMA-zeolite — subjects received boxes containing PMA-zeolite powder for supplementation for a total of 28 days.
  Dosage for PMA-zeolite (100% zeolite; 1 ML - spoon for dosage = ca. 3 g zeolite):1 spoon of the powder stirred 2 times daily (morning and evening) in water (1 glass).

SUMMARY:
The Panaceo Micro Activation (PMA) -zeolite s a certified medical device throughout the European Union and absorbs defined harmful substances (mainly heavy metals and ammonium ions) in the gastrointestinal tract, while at the same time the alkaline ions contained in the crystal lattice are released (Mg2+, Ca2+, K+, Na+). Through a recent study the main-effect of zeolite was defined (support/ strengthen the intestinal wall barrier) and as a side-effect the measurement of the mineral metabolism was included, without documenting any significant changes. Its potential in releasing minerals needs to be investigated further to broaden the knowledge from previous study-outcomes as described. Broadening this knowledge through measuring defined blood-parameters was the aim of this human trial.

DETAILED DESCRIPTION:
Background:

The ion-loaded natural PMA-zeolite do not act on the body as ion-robber in the digestive tract. The naturally occurring zeolites absorb defined ions in accordance to their selectivity alignment from their surroundings - e.g. in the gastrointestinal tract in the case of the specific certified PMA-zeolite. At the same time the PMA-zeolite absorbs defined harmful substances (mainly heavy metals and ammonium ions) in the gastrointestinal tract, while at the same time the alkaline ions contained in the crystal lattice are released (Mg2+, Ca2+, K+, Na+). Loaded with harmful substances, the zeolite is then excreted through the gastrointestinal tract without interfering with the body's metabolism.

The detoxification potential of zeolite was shown in various studies and the safety and efficacy is well documented. The measurement of the mineral metabolism was also included in a randomized controlled trial (RCT). The knowledge about its potential in releasing minerals needs however to be investigated further to broaden the knowledge from previous study-outcomes.

Methods/study-subjects:

Evaluation of the effect of the PMA-zeolite supplementation through analysis of defined blood-parameters before and after 28 days on two groups of 15 healthy volunteers (males and females) divided in NAiVE (started intake at day 1) and CHRONIC user group (intake of PMA-zeolite min. 28 before study-start).

Hypothesis:

Due to the defined effect mechanism of PMA-zeolite absorbing harmful substances (contaminants and heavy-metals) in the gastrointestinal tract and release of physiologically important minerals at the same time our hypothesis/ evaluated effects were that the PMA-zeolite has no negative impact on the mineral metabolism and might support. the natural body homeostasis, the measurement of the detoxification ability through a heavy-metal panel and other defined parameters.

Aims:

Aim of this intervention is hypothesized to lead to improvement of the enumerated values after an application after 28 days (NAiVE group).

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* at least 18 years old
* provided informed consent

Exclusion Criteria:

* chronic disease including:
* cancer,
* renal disease,
* neuro-degenerative,
* metabolic disorders,
* diabetic)
* recent vaccinations,
* pregnancy or breastfeeding,
* food supplements (if taken regularly this should be continued also during the study and documented)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Changes of Liver parameters | "Day 0" and "Day 28"
  Biochemical evaluation of LIVER PARAMETERS (aspartate-aminotransferase, alanine-aminotransferase, gamma-glutamyltransferase)
  Referent values/range used for analyses:
  aspartate aminotransferase (AST): 8-38 U/L (Unit/litre) alanine aminotransferase (ALT): 10 - 48 U/L (Unit/litre) (lower values are not clinically relevant) Gamma-glutamyl transferase (GGT): Men: 11 - 55 U/L (Unit/litre) Woman: 9 - 35 U/L (Unit/litre)
  This parameters will be combined to report the LIVER function
  The statistical analysis will be performed between this three groups of data "Changes of standard blood parameters, main standard mineral level in the blood and main metal and contaminant in the blood " , time point at "Day 0" and "Day 28" in control group and healthy volunteer group and between the groups
Changes of renal parameters | "Day 0" and "Day 28"
  Biochemical evaluation of RENAL PARAMETERS (creatinine, evaluation of the glomerular filtration speed will be done by use of a specific formula)
  Referent values/range used for analyses:
  CREAT: Woman: 63 - 107 µmol/L, Men: 79 - 125 µmol/L glomerular filtration (GF) - evaluation: G1>=90/ G2 60-80/G3a 45-59/G3b 30-40/G4 15-29/G5 <15. M: 11-32; F:8-30 µmol/l
  This parameters will be combined to report the RENAL function
  The statistical analysis will be performed between this three groups of data "Changes of standard blood parameters, main standard mineral level in the blood and main metal and contaminant in the blood " , time point at "Day 0" and "Day 28" in control group and healthy volunteer group and between the groups
Changes of main standard mineral level in the blood | "Day 0" and "Day 28"
  Evaluation of standard mineral panel
  Analyses:
  Na and K assessment relie on indirect potentiometer analysis Zn concentrations in serum assessed by use of spectrophotometric method Biochemical evaluation of Fe, Ca and Mg were done by standard spectrophotometric methods.
  Evaluation of the glomerular filtration speed will be done by use of a specific formula.
  Referent values/ range used:
  Na: 137 - 146 mmol/L; K: 3,9 - 5,1 mmol/L; Zn: Men: 11,1-19,5 μmol/l, Woman:10,7-17,5 μmol/l; Fe: Men:11-32; Woman:8-30 umol/l Mg: 0,65 - 1,05 mmol/L Ca: 2,14 - 2,53 mmol/L
  The parameters will be combined for evaluation of the mineral metabolism
  The statistical analysis will be performed between this three groups of data "Changes of standard blood parameters, main standard mineral level in the blood and main metal and contaminant in the blood " , time point at "Day 0" and "Day 28" in control group and healthy volunteer group and between the groups
Changes of main metal level in the blood | "Day 0" and "Day 28"
  Evaluation of main mineral panel
  for Pb, Hg, Cr, Cd, As, Al and Ni were inductively Coupled Plasma Mass Spectrometry-ICP-MS analysis of serum and plasma samples
  Referent values/range used:
  Lead (Pb) ≤ 50 µg/L Mercury (Hg) <10 µg/L Cadmium (Cd) < 1 µg/L Chromium (Cr) < 1 µg/L Arsenic (As) < 12µg/L Aluminium (Al) < 8 µg/L Nickel (Ni) < 2 µg/L
  The parameters will be combined for evaluation of the metal level
  The statistical analysis will be performed between this three groups of data "Changes of standard blood parameters, main standard mineral level in the blood and main metal and contaminant in the blood " , time point at "Day 0" and "Day 28" in control group and healthy volunteer group and between the groups
Changes of Meathemoglobin in the blood | "Day 0" and "Day 28"
  Methemoglobinemia is a condition of elevated methemoglobin in the blood causing headache, dizziness, shortness of breath, nausea....
  Analyses for MHgb - methaemoglobin: The method relies on CO-oximetry by use of GEM OPLTM analyser
  Referent values/range used for analyses: methaemoglobin (MHgb) : 0-1,5%
  The statistical analysis will be performed between this three groups of data "Changes of standard blood parameters, main standard mineral level in the blood and main metal and contaminant in the blood " , time point at "Day 0" and "Day 28" in control group and healthy volunteer group and between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Krešimir Pavelić, Phd, M.D., Principal Investigator — Juraj Dobrila University of Pula

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraljevic Pavelic S, Saftic Martinovic L, Simovic Medica J, Zuvic M, Perdija Z, Krpan D, Eisenwagen S, Orct T, Pavelic K. Clinical Evaluation of a Defined Zeolite-Clinoptilolite Supplementation Effect on the Selected Blood Parameters of Patients. Front Med (Lausanne). 2022 May 27;9:851782. doi: 10.3389/fmed.2022.851782. eCollection 2022. PMID 35712111